CLINICAL TRIAL: NCT02197026
Title: A Multicentre, Open-label and Randomized Clinical Trial to Compare in Patient With Knee Osteoarthritis the Medicoeconomic Benefits as Well as Effectiveness and Safety of Synvisc® Versus Usual Treatments.
Brief Title: Effectiveness and Safety of Synvisc® Versus Usual Treatments in Patients With Knee Osteoarthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1139.4
Record Dates: First submitted 2014-07-18; First posted 2014-07-22 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2014-07

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — hylan; Physical Therapy Modalities; Hydrotherapy

ARMS (2):
- Synvisc group (Experimental): injection of Synvisc® at day 1, day 8 and day 15; in the mean time it will be recommended to decrease or stop all other OA treatments
  Interventions: Drug: Hylan G-F 20
- Osteoarthritis standard treatment group (Active Comparator): Treatment will be left to the discretion of the investigator who could prescribe any therapies, except viscosupplementation product
  Interventions: Drug: Standard treatment; Procedure: Physiotherapy; Procedure: Hydrotherapy

INTERVENTIONS:
Drug: Hylan G-F 20
  Other Names: Synvisc®
  Arms: Synvisc group
Drug: Standard treatment — Standard drug treatment at the discretion of the investigator
  Arms: Osteoarthritis standard treatment group
Procedure: Physiotherapy
  Arms: Osteoarthritis standard treatment group
Procedure: Hydrotherapy
  Arms: Osteoarthritis standard treatment group

SUMMARY:
Comparison of treatment cost of knee osteoarthritis (OA) in patients treated with Synvisc® versus usual treatments as well as evaluation of safety and effectiveness of these treatments.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatient aged at least 18 years
* Patient suffering from predominant femoro-tibial knee osteoarthrosis with or without effusion. The diagnosis must be based on American College of Rheumatology (ACR) criteria. Radiological grade will be assess according to Kellgren-Lawrence scale
* Assessment of pain on active movement (i.e. walking) (by the patient) must be at least 40 mm on a 100 mm VAS
* Patient who received at least two courses of at least ten days within the last three months with non-steroidal antiinflammatory drugs (NSAID) and/or who are treated continuously for the last two month with slow-acting anti-osteoarthritis drugs
* Patient's informed written consent obtained in accordance with French legislation

Exclusion Criteria:

* Patient suffering from acute congestive osteoarthritis flare of the target knee (at the time of inclusion) which means that concomitantly to knee effusion at least 2 of the following criteria are present:

  * nocturnal disturbances due to knee pain
  * morning stiffness over 45 minutes
  * increase of knee pain more than 50% within the last week
  * articular reddening
  * articular heat
* Intra-articular administration of hyaluronic acid in the target knee within the previous year
* Intra-articular administration of hyaluronic acid in the target knee within the three previous months
* Any other intra-articular injection in the target knee within the last 6 months
* Any contraindication to intra-articular injections
* Present or past history of infected target knee joint
* Previous prosthesis knee surgery, tibial osteotomy, synovectomy or synoviorthese of the target knee
* Arthroscopy, articular lavage, debridement, menisectomy of the target knee within the previous year
* Planned knee surgery within the nine following month
* Any other musculoskeletal disorders that can interfere with osteoarthritis diagnosis or the evaluation of its severity
* Known hypersensitivity to avian products
* Presence of lymphatic or venous stasis
* Pregnancy or breastfeeding
* Clinical evidence of or known severe cardiac, hepatic, renal, metabolic, haematological disease, mental disturbance
* Participation in another clinical trial during this study or during the previous month
* Previous participation in this trial
* Patient who requires help concerning shopping or house keeping
* Patient unable to comply with the protocol (e.g. patient unable to attend each trial visit or to fill the diary booklet or the quality of life questionnaire)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 518 (Actual)
Dates: Start 1998-10; Primary Completion 2000-02 (Actual)

PRIMARY OUTCOMES:
Cost of knee OA treatment including cost of side effect related to OA treatment | up to 274 days
Area under the curve (AUC) Lequesne index | Day 1, 29, 91, 182 and 274
  Index of severity

SECONDARY OUTCOMES:
Assessment of Western Ontario and McMaster Universities (WOMAC) index by patient | Day 1, 91, 182 and 274
Patient's assessment of pain on movement and rest on a visual analogue scale (VAS) through WOMAC question 1 and 3 | Day 1, 91, 182 and 274
Disease activity assessment by patient and investigator on a VAS | Day 1, 29, 91, 182 and 274
Acute congestive OA flares assessed through a questionnaire | Day 1, 29, 91, 182 and 274
Assessment of state of health of the patients with a quality of life questionnaire (SF 12) | Day 1, 91, 182, 274
Final global assessment of efficacy by patient and investigator on a four-point verbal rating scale (VRS) | Day 274
Final global assessment of tolerability by patient and investigator on a four-point VRS | Day 274
Incidence and intensity of adverse events | up to day 274
Number of withdrawals due to adverse event | up to day 274